CLINICAL TRIAL: NCT03178825
Title: Safety and Efficacy of Hybrid Fractional Laser Treatment for Symptoms of Genitourinary Syndrome of Menopause
Brief Title: Hybrid Fractional Laser for Symptoms of Genitourinary Syndrome of Menopause
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sciton (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIVACIP002
Record Dates: First submitted 2017-06-05; First posted 2017-06-07 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Vaginal Atrophy; Sexual Dysfunction; Dyspareunia; Vaginal Dryness; Chronic UTI
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Dyspareunia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Hybrid Fractional Laser (Experimental): Hybrid fractional 2940 nm and 1470 nm laser treatment
  Interventions: Device: Hybrid Fractional Laser

INTERVENTIONS:
Device: Hybrid Fractional Laser — Consecutive and coincident fractional 2940 nm and 1470 nm lasers
  Other Names: diVa

SUMMARY:
This multi-center clinical trial will evaluate the safety and long-term efficacy of hybrid fractional 2940 nm and 1470 nm lasers for treatment of symptoms of Genitourinary Syndrome of Menopause.

DETAILED DESCRIPTION:
Both 2940 nm Er:YAG (Erbium-doped yttrium aluminium garnet) and 1470 nm diode lasers are cleared by the Food and Drug Administration (FDA) for ablation, vaporization, coagulation of soft tissue and for skin resurfacing. Fractional delivery of laser is a well-established method that stimulates tissue remodeling in the dermis while leaving the surrounding tissue intact in order to decrease healing time. The layers of skin and vaginal mucosal tissue exhibit similarities that suggest the clinical results seen with skin resurfacing may be translated to the vaginal tissue. Improved vaginal tissue health may lead to improvement of symptoms of Genitourinary Syndrome of Menopause (GSM). This multi-centered, 18-month prospective clinical trial will evaluate the safety and long-term effectiveness of hybrid fractional 2940 nm and 1470 nm lasers (HFL) as an alternative non-surgical, non-hormonal treatment for symptoms of GSM.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy biological female aged between 40 to 70 years
2. Is post-menopausal with a AND b OR c

   1. No menses for at least 12 months
   2. Follicle-stimulating hormone (FSH) level over 40mlU/mL
   3. Has had a bilateral oophorectomy at least 12 months ago with no hormone replacement
3. Is experiencing at least two self-reported symptoms of GSM, such as

   1. Vaginal irritation in absence of infection
   2. Chronic burning sensation
   3. Chronic itching in the absence of infection
   4. Recurring urinary tract infections (UTIs)
   5. Vaginal dryness during sexual activity
   6. Pain during sexual activity (dyspareunia)
4. Has been experiencing symptoms of GSM for greater than 3 months
5. Is unable due to medical contraindication or unwilling to receive hormone-based vaginal therapy
6. Normal and up-to-date pap smear if applicable
7. Is sexually active (i.e. intravaginal intercourse) or has the potential and desire to be sexually active if symptoms of GSM improve
8. Can read, understand and sign informed consent form

Exclusion Criteria:

1. Undiagnosed abnormal genital bleeding
2. Has history of pelvic surgery or other energy-based vaginal therapy within 6 months prior to enrollment
3. Previous use of topical estrogen therapy within the last 3 months
4. Has used vaginal creams, moisturizers, lubricants or homeopathic preparations or received anticoagulants, antiplatelet, thrombolytic, vitamin E or anti-inflammatory within 2 weeks of treatment
5. History of heart failure
6. Has equal to or greater than stage III prolapse, according to pelvic organ prolapse quantification system (POP-Q)
7. Has an active sexually transmitted infection (STI)
8. Has signs or symptoms of vaginitis/vulvitis
9. Has signs or symptoms of acute urinary tract infection (UTI)
10. Has participated in any clinical trial involving an investigational drug or procedure within the past 30 days
11. The investigator feels that for any reason the subject is not eligible to participate in the study

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal Females
Enrollment: 60 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Vaginal Maturation Index (VMI) | 12 months
  An objective assessment of vaginal hormone response as well as overall hormonal environment by calculating a ratio of parabasal cells, intermediate cells, and superficial cells

SECONDARY OUTCOMES:
Change from baseline in Histology | 12 months
  Change from baseline in epithelial thickness, collagen, elastin, vascularity, and fibroblast density.
Change from baseline in Vaginal Health Index Score (VHIS) | 12 months
  A quantitative assessment of vaginal health that evaluates vaginal elasticity, fluid volume, pH, epithelial integrity, and moisture on a scale of 1 to 5.
Change from baseline in Female Sexual Function Index (FSFI) | 12 months
  A multidimensional self-report instrument for assessment of female sexual function.
Change from baseline in Day-to-Day Impact of Vaginal Aging Questionnaire (DIVA) | 12 months
  A multidimensional self-report measure of the impact of vaginal symptoms on functioning and well-being in postmenopausal women.
Change from baseline in Clinical Photography | 12 months
  Change from baseline in the appearance of the treatment area.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Guerette, MD, Principal Investigator — The Female Pelvic Institute of Virginia
Locations (6):
- United States (6):
  - Women's Pelvic Health Institute, Los Gatos, California
  - Coyle Institute, Pensacola, Florida
  - Louisiana State University, New Orleans, Louisiana
  - Carolinas Healthcare System, Charlotte, North Carolina
  - Woodlands Gynecology & Aesthetics, The Woodlands, Texas
  - The Female Pelvic Medicine Institute of Virginia, North Chesterfield, Virginia

IPD SHARING:
Plan to Share IPD: No